CLINICAL TRIAL: NCT06528860
Title: The Effectiveness and Acceptability of Dual-focus Soft Contact Lenses for Controlling Rapid Progressive Myopia in Young Adults: A Randomized Controlled Trial
Brief Title: Dual-focus Soft Contact Lenses for Controlling Rapid Progressive Myopia in Young Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QX-2024-A-002
Record Dates: First submitted 2024-07-26; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Myopia
Keywords: Myopia; Dual-focus contact lenses; Young adults; Adult myopia progression
MeSH Terms: conditions — Myopia | interventions — Contact Lenses, Hydrophilic

STUDY DESIGN:
Intervention Model Description: Intervention Group: Daily disposable bifocal soft corneal contact lenses: MiSight® 1 day soft contact lens (CooperVision, material: omafilcon A, water content: 60%).
  Control Group: Daily disposable single-focus soft corneal contact lenses: Proclear® 1 day soft contact lens (CooperVision, material: omafilcon A, water content: 60%)
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study will utilize a Central Randomization System (CRS) for the random grouping and glasses allocation of study subjects during the clinical trial. Investigators and participants will be blinded to the intervention received until unblinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual-focus CL (Experimental): Wearing dual-focus CL for 2 years
  Interventions: Device: MiSight® 1 day soft contact lenses
- Single-vision CL (Placebo Comparator): Wearing single-vision CL for 2 years
  Interventions: Device: Proclear® 1 day soft contact lenses

INTERVENTIONS:
Device: MiSight® 1 day soft contact lenses — Dual-focus contact lenses, daily disposable, material: omafilcon A, water content: 60%.
  Other Names: CooperVision
  Arms: Dual-focus CL
Device: Proclear® 1 day soft contact lenses — Single-vision contact lenses, daily disposable, material: omafilcon A, water content: 60%.
  Other Names: CooperVision
  Arms: Single-vision CL

SUMMARY:
This study aims to evaluate the effectiveness and acceptability of dual-focus soft contact lenses in controlling rapid myopia progression in adults through a randomized controlled trial. By applying myopia control measures to the adult population, we hope to provide scientific evidence for the effective control of adult myopia progression and offer insights into the understanding of myopia progression during early adulthood.

DETAILED DESCRIPTION:
It has long been believed that the progression of myopia mainly occurs during the elementary to high school stages. However, some studies and clinical practice suggest that a considerable proportion of adults still experience myopia progression in their adulthood, especially in those who have prolonged near work or screen usage time. At present, there is insufficient evidence on whether these population needs myopia control intervention. Most adults experiencing myopia progression do not receive appropriate myopic intervention measures, leading to an increase of dioptre, which may affect the quality of daily life, and raise the risk of high myopia and blinding myopia complications.

This study aims to evaluate the effectiveness and acceptability of dual-focus soft contact lenses in controlling rapid myopia progression in adults through a randomized controlled trial. By applying myopia control measures to the adult population, we hope to provide scientific evidence for the effective control of adult myopia progression and offer insights into the understanding of myopia progression during early adulthood.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-25 years;
* Myopia progression <= -0.50D in either eye in the past year (evaluated by -manifest refraction);
* The subject eye: cycloplegic spherical equivalent ranges from -2.00D to -6.0D and cylinder power doesn't exceed -1.50D;
* The subject eye's best corrected visual acuity <= logMAR 0.1;
* Anisometropia does not exceed 1.50D.

Exclusion Criteria:

* Current use of MC interventions or prior use of MC interventions within the past 6 months;
* Disease or anatomical factors that affect the wearing of contact lenses;
* History of myopia correction surgery;
* Suffering from ocular or systemic diseases that may be related to myopia, such as Marfan syndrome, retinopathy of prematurity, diabetes, etc.;
* pregnant female;
* Other conditions deemed unsuitable by the investigators.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-08-31 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in cycloplegic spherical equivalent after 2 years | 2 years after the baseline
  The difference in the change of cycloplegic spherical equivalent between the intervention group and the control group.

SECONDARY OUTCOMES:
Change in axial length after 2 years | 2 years after the baseline
  The difference in the change of axial length between the intervention group and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangui He, Principal Investigator — Shanghai Eye Disease Prevention & Treatment Center
Locations (1):
- Shanghai Eye Disease Prevention & Treatment Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruiz-Pomeda A, Villa-Collar C. Slowing the Progression of Myopia in Children with the MiSight Contact Lens: A Narrative Review of the Evidence. Ophthalmol Ther. 2020 Dec;9(4):783-795. doi: 10.1007/s40123-020-00298-y. Epub 2020 Sep 11. PMID 32915454
- [Background] Bullimore MA, Lee SS, Schmid KL, Rozema JJ, Leveziel N, Mallen EAH, Jacobsen N, Iribarren R, Verkicharla PK, Polling JR, Chamberlain P. IMI-Onset and Progression of Myopia in Young Adults. Invest Ophthalmol Vis Sci. 2023 May 1;64(6):2. doi: 10.1167/iovs.64.6.2. PMID 37126362